CLINICAL TRIAL: NCT03263676
Title: Randomized Controlled Crossover Comparison of Icon Underwear to Disposable Pads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-042
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Reusable Underwear, Urinary Incontinence, Dispoable Pad
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icon reusable underwear (Experimental)
  Interventions: Device: Disposable pad
- Disposable pad (Placebo Comparator)
  Interventions: Device: Icon resuable underwear

INTERVENTIONS:
Device: Icon resuable underwear — Reusable incontinence underwear
  Arms: Disposable pad
Device: Disposable pad — Standard market disposable pad
  Arms: Icon reusable underwear

SUMMARY:
This is a randomized cross over trial to compare quality of life and product performance between Icon reusable underwear versus standard disposable pad in patients with mild to moderate urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence is estimated to affect approximately 1/5 of all women in the United States. Multiple studies have compared effectiveness, cost-effectiveness and comfort of a variety absorbent products but most of the current data compares daily disposable insert pads. Icon reusable underwear is a new product on the market for light incontinence (25-30mL daily). The primary objective of this randomized cross over trial is to compare quality of life and patient comfort and to determine patient preference using Icon reusable underwear versus standard incontinence pad in the management of urinary incontinence. The secondary objective is to compare the cost-effectiveness of ICON underwear to disposable pads. Women with small to moderate urinary incontinence to use either ICON underwear or pads for two days and then crossed over to use other product for two days. The primary outcome measures were Incontinence Quality of Life Instrument 3 (I-QOL) and Product Performance Questionnaire 4 (PPQ) after use of each product. A sample size of 70 was calculated to detect a difference of 10.0 in the I-QOL to achieve a power of 80% with a significance level of 0.05 and to account for a 20% attrition.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are at least 18yo
* Mild to moderate urinary incontinence, defined as a response "small" or "moderate" amount to the ICIQ-SF question - "How much do you leak?"

Exclusion Criteria:

* Active urinary tract infection
* Fecal incontinence, defined as a response "large" amount to the ICIQ-SF question - "How much do you leak?"

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Incontinence Quality of Life Questionnaire | 2 days
  Validated quality of life questionnaire

SECONDARY OUTCOMES:
Product Performance Questionnaire | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Lee Richter, Principal Investigator — Medstar Health Research Institute

IPD SHARING:
Plan to Share IPD: Undecided